CLINICAL TRIAL: NCT06878235
Title: Validation of the French Version of the PLSFRS Scale
Brief Title: Validation of the French Version of the Primary Lateral Sclerosis Functioning Rating Scale (PLSFRS)
Acronym: FRENPRILS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240260-FRENPRILS
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lateral Sclerosis
Keywords: Scale
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a primary lateral sclerosis
  Interventions: Other: Assessment of the functional status

INTERVENTIONS:
Other: Assessment of the functional status — assessment of their functional status using the French version of the PLSFRS scale during a routine multidisciplinary assessment every 3-6 months for all patients with motor neurone disease, as recommended by the FILSLAN network

SUMMARY:
This is a national, multicentric, prospective, descriptive study evaluating the psychometric properties of the French version PLSFRS scale

DETAILED DESCRIPTION:
This is a prospective study conducted in 8 French ALS centers which will enroll 80 patients with PLS. All these patients will undergo an evaluation of their functional status from the ALSFRS-r and PLSFRS scales. All patients will be evaluated at 3 time points (T0,M6 at the outpatient clinic) and at M3 remotely. The aim of the study will be to validate a trans-cultural and psychometric version of the PLSFRS available for the French PLS population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary lateral sclerosis (PLS)
* Age over 18 years
* Informed consent signed
* Patients cared in a French ALS centre

Exclusion Criteria:

* patients with no oral and written command of the French language
* Patients unable to answer a questionnaire
* Opposition to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary lateral sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
French version of the PLSFRS scale | inclusion and 6 months
  10 items with a score from 0 to 6; 2 items with a score from 0 to 4 Maximal score is 68.

SECONDARY OUTCOMES:
Change Global Impression (CGI) scale | 6 months
  overall clinical impression of the change; score from 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CORCIA, PR, Principal Investigator — University Hospital, Tours
Locations (7):
- France (7):
  - University hospital, Brest
  - University hospital, Clermont-Ferrand
  - University hospital, Lille
  - University hospital, Limoges
  - University hospital, Lyon
  - University Hospital, Nice
  - University hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided